CLINICAL TRIAL: NCT06208774
Title: Pericapsular Nerve Group Block vs Low Volume Interscalene Brachial Plexus Block for Shoulder Arthroscopy: A Randomized Controlled Trial
Brief Title: Pericapsular Nerve Group Block vs Interscalene Block for Shoulder Arthroscopy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nagy Malak , MD, Lecturer anesthesia cairo university, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: N-403-2023
Record Dates: First submitted 2023-12-09; First posted 2024-01-17 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Anesthesia; Regional Anesthesia Morbidity; Shoulder Pain; Arthroscopy
Keywords: Shoulder; PENG; Interscalene block; Arthroscopy
MeSH Terms: conditions — Shoulder Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LV-ISBP block Group (n=40): US-guided low volume interscalene brachial plexus block (Experimental): Patient in a semi-sitting position with the head tilted to the opposite side of the injection site. A linear US probe (4-12 MHz) will be placed parallel to the clavicle in the supraclavicular fossa, and the subclavian artery will be seen beating above the first rib.Then the probe will be moved cranially to identify the transverse process of the C7 vertebra at the level of the brachial plexus roots between the scalenus anterior and medius muscles.The needle will be inserted in a plane approach from lateral to medial to scalenus medius and C5-C6 brachial plexus roots. After negative aspiration, a total of 5 mL of bupivacaine 0.5% will be injected incrementally.
  Interventions: Procedure: Ultrasound-guided PENG or ISBP block
- PENG block Group (n=40): US-guided pericapsular nerve group block for shoulder (Active Comparator): The patient's arm was placed in external rotation and abducted at 45 degrees. A linear US probe (4-12 MHz) will be placed longitudinally between the coracoid and the humeral head, visualizing the deltoid muscle and subscapularis tendon. 22-gauge needle will be advanced in-plane into the fascial plane between the deltoid muscle and subscapularis tendon. The location of the needle tip will be confirmed by hydrodissection of inter-fascial planes with 3 ml of normal saline. After negative aspiration, a total of 20 mL of bupivacaine 0.5% will be injected in the fascial plane incrementally, aspirating every 5 ml.
  Interventions: Procedure: Ultrasound-guided PENG or ISBP block

INTERVENTIONS:
Procedure: Ultrasound-guided PENG or ISBP block — The diaphragmatic excursion will be measured in the supine position before the block and after surgery. A curvilinear US probe (5-7 MHz) will be placed at the subcostal area in the anterior axillary line, below the costal margin of the eighth and ninth ribs. The probe will be directed medially, cephalad, and dorsally to make the US beam reach the posterior third of the diaphragm perpendicularly. The probe will then be scanned along the long axis of the intercostal spaces, using the liver as the acoustic window on the right side and the spleen as on the left side. M-mode sampling line will be positioned perpendicularly to the diaphragm, and the diaphragmatic excursions could be measured during quiet and deep breathing.The measurement will be repeated three times, and the average value will be taken. After measurement of diaphragmatic excursion, patients will receive either a PENG block or an LV-ISBP block before induction of general anesthesia.

SUMMARY:
This study aims to compare PENG block and LV-ISBP block in the incidence of phrenic nerve block, duration of postoperative analgesia, time to first analgesic request (VAS > 30 mm), pain scores, and side effects.

DETAILED DESCRIPTION:
This randomized, controlled, double-blinded trial will be conducted in a Cairo University hospital.On arrival of the patients in the regional anesthesia room, they will be secured with a 20-gauge intravenous cannula. Monitoring will include ECG, non-invasive arterial blood pressure, and pulse oximetry (SpO2).

Before receiving the blocks, patients will be randomly assigned to one of the two study groups for diaphragmatic movement assessment:

The diaphragmatic excursion will be measured in the supine position before the block and after surgery by a blinded operator. A curvilinear ultrasound probe (5-7 MHz) will be placed at the subcostal area in the anterior axillary line, below the costal margin of the eighth and ninth ribs. The probe will be directed medially, cephalad, and dorsally to make the ultrasound beam reach the posterior third of the diaphragm perpendicularly. The probe will then be scanned along the long axis of the intercostal spaces, using the liver as the acoustic window on the right side and the spleen as the acoustic window on the left side. The M-mode sampling line will be positioned perpendicularly to the diaphragm, and the diaphragmatic excursions could be measured during quiet and deep breathing. The distance between the resting expiratory position and the maximum deep inspiration position will be measured. The measurement will be repeated three times, and the average value will be taken.

After measurement of diaphragmatic excursion, patients will receive either a PENG block or an LV-ISBP block before induction of general anesthesia, and to achieve double blinding, patients will receive the block by consultant anesthesiologists who have experience in regional anesthesia. Another doctor not involved in the block procedure will evaluate the patient intraoperatively and postoperatively.

PENG block group (n = 40): this group will receive an ultrasound-guided pericapsular nerve group block for the shoulder with a total volume of 20 mL and 0.5% bupivacaine.

LV-ISBP block group (n = 40): this group will receive ultrasound-guided low-volume interscalene brachial plexus block with a total volume of 5 mL and 0.5% bupivacaine.

Technique of PENG Block:

The technique of ultrasound-guided PENG block will be performed with the patient's arm placed in external rotation and abducted at 45 degrees. A linear ultrasound probe (4-12 MHz) will be placed longitudinally between the coracoid and the humeral head, visualizing the deltoid muscle and subscapularis tendon. A 22-gauge needle will be advanced in-plane, into the fascial plane between the deltoid muscle and subscapularis tendon. The location of the needle tip will be confirmed by hydrodissection of inter-fascial planes with 3 ml of normal saline. After negative aspiration, a total of 20 mL of bupivacaine 0.5% will be injected in the fascial plane incrementally, aspirating every 5 ml.

Technique of the LV-ISBP block:

The technique of ultrasound-guided LV-ISBP will be performed with the patient in a semi-sitting position with the head tilted to the opposite side of the injection site. A linear ultrasound probe (4-12 MHz) will be placed parallel to the clavicle in the supraclavicular fossa, and the subclavian artery will be seen beating above the first rib. Then the probe will be moved cranially to identify the transverse process of the C7 vertebra at the level of the brachial plexus roots between the scalenus anterior and medius muscles. A volume of 2 mL of 2% lignocaine will be infiltrated subcutaneously before the block. The needle will be inserted in a plane approach from lateral to medial to scalenus medius and C5-C6 brachial plexus roots. The location of the needle tip will be confirmed by hydrodissection with 1 ml of normal saline. After negative aspiration, a total of 5 mL of bupivacaine 0.5% will be injected incrementally, aspirating every 2.5 mL.

To ensure blind assessment, a dressing will be placed to cover a standard area that will cover the puncture sites regardless of which block is performed.

In the operating room, induction of general anesthesia will be induced after adequate preoxygenation using 1 µg/kg fentanyl, 2 mg/kg propofol, and 0.5 mg/kg atracurium, in addition to 8mg IV dexamethasone for the prevention of postoperative nausea and vomiting. Endotracheal intubation will be established. Anesthesia will be maintained by 1.2% MAC of isoflurane with oxygen (50%) in the air, and 0.1 mg/kg of atracurium will be administered every 20 minutes as maintenance anesthetic drugs. Volume-controlled ventilation will be maintained, and the respiratory rate will be adapted to maintain ET CO2 between 35 and 40 mmHg. Monitoring through ECG, NIBP, pulse oximetry, and capnography (ETCO2) continued throughout the surgeries. Each portal skin of the arthroscopy will be infiltrated by the surgeon with approximately 4 mL of 0.25% bupivacaine. Intraoperative inadequate analgesia, indicated by an increase in HR or mean arterial blood pressure (MAP) more than 20% above preinduction baseline values, will be managed using incremental 50-microgram doses of fentanyl. Intraoperative fentanyl consumption will be calculated. All patients will receive ketorolac 30mg IV and paracetamol 1 mg for postoperative analgesia. At the end of surgery, muscle relaxants will be reversed using neostigmine 0.05 mg/kg and atropine 0.02 mg/kg. Awake extubation will be established after adequate reversal of the neuromuscular block.

Patients will be transported to the post-anesthesia care unit (PACU) for one hour before being shifted to the ward. In the PACU, after the patient regains full consciousness, the diaphragmatic movement will be reassessed in the exact same manner as preoperatively. Phrenic nerve block is defined as failure of the diaphragm to achieve 25% of the pre-block excursion value.

Postoperative pain will be assessed using VAS (where 0 corresponds to no pain and 100 mm to the worst pain) at 2, 4, 6, 12, 18, and 24 hours postoperatively.

Postoperatively, in the ward, all patients will receive 1 g paracetamol every 6 h and 30 mg ketorolac every 12 h. If the VAS score is > 30 mm, IV morphine increments (2 mg) will be given to maintain VAS ≤ 30 mm with a maximum total 24-hour morphine consumption of 10 mg, and total morphine consumption will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for shoulder arthroscopy
* American Society of Anesthesiologists (ASA) status I and II
* Ages between 18 and 60 years.

Exclusion Criteria:

* Coagulopathy
* Infection at the injection site.
* Allergy to local anesthetics
* Severe cardiopulmonary disease (≥ASA III)
* Diabetic or other neuropathies
* Motor disorders
* Patients receiving opioids for chronic analgesic therapy.
* Inability to comprehend visual analogue scale (VAS).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-12-20 (Actual); Primary Completion 2024-05-30 (Estimated); Study Completion 2024-05-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of phrenic nerve block | 24 hours
  Incidence of phrenic nerve block

SECONDARY OUTCOMES:
First analgesic request | 24 hours postoperative
  Time to first analgesic request (Visual analogue pain> 40 mm)
Visual analogue pain score | 24 hours postoperatively.
  Visual analogue pain score for pain assessment (from 0 the Best to 100 the worst) at 2, 4, 6, 12, 18, and 24 hours postoperatively
Total morphine requirements | 24 hours
  Total morphine requirements 24 hours postoperatively.
Type and time of surgery | up to 4 hours
  Type and time of surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo university Hospitals. kasralainy, Cairo, Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided